CLINICAL TRIAL: NCT07105852
Title: Exploring the Safety and Efficacy of Sacituzumab Tirumotecan Combined With Pucotenlimab in the Treatment of Advanced Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRRSH2025-0390
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First-line treatment cohort for advanced cholangiocarcinoma (Not treated before) (Active Comparator): Intervention:Sacituzumab tirumotecan (iv)+Putolizumab injection (iv)
  Interventions: Drug: Sacituzumab tirumotecan (iv)+Putolizumab injection (iv)
- Second-line treatment cohort for advanced cholangiocarcinoma (Treated before, but failed) (Experimental): Intervention:Sacituzumab tirumotecan (iv)+Putolizumab injection (iv)
  Interventions: Drug: Sacituzumab tirumotecan (iv)+Putolizumab injection (iv)

INTERVENTIONS:
Drug: Sacituzumab tirumotecan (iv)+Putolizumab injection (iv) — When administering sacituzumab tirumotecan and putolizumab on the same day, the drugs should be given sequentially. Putolizumab is administered first. For the first co-administration, a 4-hour interval is required. If no severe infusion reactions or allergic reactions occur, subsequent administrations may proceed with a minimum interval of 60 minutes before administering sacituzumab tirumotecan.
  Putolizumab dosing:
  Dosage: 200 mg, intravenous (IV) infusion Dosing cycle: Every 3 weeks (administered on Day 1 of each cycle) Dose interruptions due to adverse events (AEs): Refer to the prescribing information.
  Sacituzumab tirumotecan dosing:
  Dosage: 4 mg/kg, intravenous (IV) infusion Dosing cycle: Every 2 weeks (administered on Day 1 of each cycle, with a permissible dosing window of 14 ± 3 days between doses) Dose interruptions due to adverse events (AEs): Refer to the prescribing information.

SUMMARY:
1. Primary Objectives (1) To evaluate the safety and tolerability of sacituzumab tirumotecan in combination with pucotenlimab in patients with advanced cholangiocarcinoma; (2) To assess the objective response rate (ORR) of sacituzumab tirumotecan combined with pucotenlimab in patients with unresectable or metastatic cholangiocarcinoma, as evaluated by investigators per RECIST v1.1;
2. Secondary Objectives (1) To evaluate the overall survival (OS) of sacituzumab tirumotecan combined with pucotenlimab in advanced cholangiocarcinoma; (2) To assess progression-free survival (PFS), disease control rate (DCR), duration of response (DOR), and time to response (TTR) in patients treated with sacituzumab tirumotecan combined with pucotenlimab, as determined by investigators based on RECIST v1.1; (3) To further evaluate PFS (as a standalone secondary endpoint);
3. Exploratory Objectives (1) To investigate the correlation between TROP2 expression, systemic immune biomarkers, and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >= 18 years old; 2. Histologically confirmed unresectable or metastatic cholangiocarcinoma (including gallbladder cancer, intrahepatic cholangiocarcinoma, and extrahepatic cholangiocarcinoma)

  (1) First line treatment cohort:
  1. Patients who explicitly refuse chemotherapy;
  2. Patients who fail adjuvant therapy with chemotherapy;
  3. Patients who have not received systemic therapy; (2) Second line treatment cohort:

  <!-- -->

  1. First line chemotherapy is effective, but toxicity is not tolerated;
  2. Disease progression after first-line chemotherapy regimen]; 3. Patients with positive TROP2 protein; 4. The patient is a patient with distant metastasis or locally advanced stage who cannot undergo surgery or radiotherapy and has not received systemic treatment; 5. According to RECIST 1.1 tumor evaluation criteria, there is a measurable primary lesion; 6. No active autoimmune diseases; 7. No concurrent malignant tumors; 8. ECOG physical fitness score 0-1; 9. Expected survival period >= 3 months; 10. Having sufficient organ and bone marrow function (not receiving blood transfusions, recombinant human thrombopoietin or colony-stimulating factor therapy within 2 weeks prior to the first administration), defined as follows:

  <!-- -->

  1. Blood routine: neutrophil count (NEUT) >= 1.2 × 10^9/L; platelet count (PLT) >= 75 × 10^9/L; hemoglobin >= 9 g/dL;
  2. Liver function: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) <= 2.5 x upper limit of normal (ULN); Total bilirubin (TBIL) <= 1.5 × ULN; If there is liver metastasis, ALT and AST should be <= 5ULN;
  3. Renal function: plasma Cr <= 1.5ULN or creatinine clearance rate (Ccr) >= 60 ml/min (for males: GFR (ml/min)=(140 age) x body weight (kg) x 0.85/blood creatinine (mg/dl); For women: GFR (ml/min)=(140 age) x body weight (kg) x 0.85 x 0.85/blood creatinine (mg/dl);
  4. Coagulation function: International normalized ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) <= 1.5 × ULN; 11. For female subjects with fertility and male subjects with reproductive potential partners, they must agree to take effective medical contraceptive measures within 6 months from the signing of the informed consent form until the last administration; 12. Voluntarily join this study and sign an informed consent form. If the subject is unable to read and sign the informed consent form due to reasons such as lack of capacity, their guardian needs to act as a proxy for the informed process and sign the informed consent form. If the subject lacks the ability to read the informed consent form (such as illiterate subjects), a witness is required to witness the informed process and sign the informed consent form.

     Exclusion Criteria:
* 1. Previously received any of the following treatments (including in the context of adjuvant or neoadjuvant therapy): targeted TROP2 therapy; Any drug therapy containing targeted topoisomerase I, including antibody conjugated drug (ADC) therapy; Immune checkpoint inhibitors (such as anti-PD-1/L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immune cell therapy, and any other treatment targeting the tumor immune mechanism; 2. Suffering from other malignant tumors within 3 years before administration (excluding tumors that have been cured through local treatment, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, cervical carcinoma in situ, etc.); 3. Ampullary cancer; 4. Previously received ADC targeting TROP2 or any drug treatment containing topoisomerase I inhibitors; 5. Allergies to any components of the investigational drugs (sacituzumab tirumotecan and pucotenlimab); 6. There is a history of (non infectious) interstitial lung disease (ILD) or non infectious pneumonia that requires steroid treatment, current ILD or non infectious pneumonia, or suspected ILD or non infectious pneumonia that cannot be excluded by imaging examination during screening; 7. Suffering from active autoimmune diseases that require systematic treatment within the past two years (including but not limited to: autoimmune hepatitis, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, etc.). Hormone replacement therapy, such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered systemic therapy; 8. Any disease requiring systemic corticosteroid treatment (dose>10 mg/d of prednisolone or equivalent dose of similar drugs) or other immunosuppressive therapy within 10 days prior to the first study treatment. However, subjects who receive intranasal, inhaled, topical, or local corticosteroid injections (such as intra-articular injections), or corticosteroids as a preventive medication for hypersensitivity reactions, may be included; 9. Known active pulmonary tuberculosis. Subjects suspected of having active pulmonary tuberculosis need to undergo clinical examination for exclusion; 10. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation; 11. Diagnosed as active hepatitis B or C; 12. Human immunodeficiency virus (HIV) test is positive or there is a history of acquired immunodeficiency syndrome (AIDS); Known active syphilis infection; 13. Suffering from local or systemic diseases caused by non malignant tumors, or diseases or symptoms secondary to tumors, which can lead to higher medical risks and/or uncertainty in survival evaluation, such as tumor like leukemia reactions, cachexia manifestations, etc.; 14. There is a recorded history of severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or corneal diseases that hinder/delay corneal healing; 15. Unable to comply with the visit and related procedures stipulated in the plan; 16. Pregnant or lactating women; 17. Vulnerable groups other than the elderly/illiterate, including critically ill patients, individuals with mental illnesses, and those with cognitive impairments; 18. The researcher believes that the patient is not suitable to participate in any other circumstances of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 year

SECONDARY OUTCOMES:
Overall survival (OS) | 2 year
Disease control rate (DCR) | 2year
Progression-free survival (PFS) | 2 year
Duration of response (DOR) | 2 year

OTHER OUTCOMES:
The incidence, severity, and correlation with the investigational product of adverse events (all adverse events, treatment emergent adverse events, serious adverse event) | 2 year
Biomarkers (TROP2 protein detection, CA-199, AFP, CEA) | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine (Qingchun Campus) 3 Qingchun Road East, Shangcheng District, Hangzhou, Zhejiang, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No